CLINICAL TRIAL: NCT01090999
Title: Long - Term Respiratory Rehabilitation Programs in Chronic Obstructive Pulmonary Disease (COPD) Patients: Study of Cost- Effectiveness.
Brief Title: Long - Term Respiratory Rehabilitation Programs in Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR04/04/2007
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): All patients will receive an initial in-hospital rehabilitation program which includes: Education, Physiotherapy, lower and upper extremities training and respiratory muscles training. Following completion of this program, patients will undergo concealed randomization to one of two maintenance strategies.
  The No Intervention group will undergo a standard, minimal monitoring program.
- 2 (Active Comparator): All patients will receive an initial in-hospital rehabilitation program which includes: Education, Physiotherapy, lower and upper extremities training and respiratory muscles training. Following completion of this program, patients will undergo concealed randomization to one of two maintenance strategies.
  The active comparator group will undergo an intensive maintenance program after the initial in-hospital rehabilitation program.
  Interventions: Other: long-term maintenance respiratory rehabilitation program

INTERVENTIONS:
Other: long-term maintenance respiratory rehabilitation program — To determine whether a long-term maintenance program after respiratory rehabilitation (group active comparator), in contrast to the usual minimal maintenance therapy (group no intervention), improves the cost-effectiveness through: a.- maintaining long term effects in terms of effort capacity, HRQL, and reduced exacerbations b.- reducing the total cost of care to patients, largely through reduction of exacerbations.
  Arms: 2

SUMMARY:
OBJECTIVE: To determine whether a long-term maintenance program after respiratory rehabilitation, in contrast to the usual minimal maintenance therapy, improves the cost-effectiveness through: a.- maintaining long term effects in terms of effort capacity, HRQL, and reduced exacerbations b.- reducing the total cost of care to patients, largely through reduction of exacerbations.

MATERIAL AND METHODS: multi-center (4 hospitals) prospective randomized controlled study that will include 150 patients with moderate-severe COPD (age <75; BODE 4-10) with a 3 years follow-up. All patients will receive an initial in-hospital rehabilitation program which includes: Education, Physiotherapy, lower and upper extremities training and respiratory muscles training. Following completion of this program, patients will undergo concealed randomization to one of two maintenance strategies:1.-an intensive maintenance program (GR1) 2.- a standard, minimal monitoring program (GR2). On the intensive maintenance program (GR1) the physiotherapist will call once a week as a reminder and the patient will attend the hospital once a week . A physiotherapist will supervise the weekly in-hospital exercise and he/she will check if the patient is properly undergoing the rehabilitation treatment.

OUTCOMES: 1.- Clinical: dyspnea (area of CRQ questionnaire), HRQL (CRQ, SF 36); Effort capacity (6minute Walking Test), BODE index; 2.- Economical: direct costs (programs); indirect costs (exacerbations, admissions); comparison of GR1 and GR2 costs; EXPECTED OUTCOMES: reduction of dyspnea, improvement of HRQL, effort capacity and BODE index, and reduction of health expenditures in GR1 compared to GR2.

ELIGIBILITY:
Inclusion Criteria:

* COPD Patients
* Less than 77 years
* BODE index of 3-10 (BODE 3 when FEV1<50% v. Ref.).
* clinically stable (at least one month)
* Informed consent signed

Exclusion Criteria:

* Bone or muscle disease that limits the exercise training.
* Heart disease that disable physic exercise.
* Bronchiectasis or other Respiratory diseases different than COPD.
* Comorbidity that difficult o disable respiratory rehabilitation program carrying out.
* Life expectation less than 2 years.

Max Age: 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
1.- Clinical: dyspnea (area of CRQ questionnaire), | 1.5 YEARS
Effort capacity (6minute Walking Test), | 1.5 Years
BODE index; | 1.5 Years
Economical: direct costs (programs); | 1.5 Years
indirect costs (exacerbations, admissions); | 1.5 Years
comparison of GR1 and GR2 costs; | 1.5 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Guell MR, Cejudo P, Ortega F, Puy MC, Rodriguez-Trigo G, Pijoan JI, Martinez-Indart L, Gorostiza A, Bdeir K, Celli B, Galdiz JB. Benefits of Long-Term Pulmonary Rehabilitation Maintenance Program in Patients with Severe Chronic Obstructive Pulmonary Disease. Three-Year Follow-up. Am J Respir Crit Care Med. 2017 Mar 1;195(5):622-629. doi: 10.1164/rccm.201603-0602OC. PMID 27611807